CLINICAL TRIAL: NCT06890637
Title: Efficacy of Microbiome Manipulation Strategies (Fecal Microbial Transplant or Crohns Disease Exclusion Diet or Both) With Advanced Therapies (BiOlOgics and Small Molecules) to Break the Therapeutic Ceiling in Active Crohns Disease (BOOST-CD): A Multicenter Double Blind Factorial Randomized Controlled Trial
Brief Title: A Study to Evaluate the Effect of Fecal Transplant and Dietary Changes on Disease Activity in Patients With Crohn Disease on Advanced Therapies
Acronym: BOOST-CD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Prof. Vineet Ahuja, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMSA2988/03.01.2025
Record Dates: First submitted 2025-03-03; First posted 2025-03-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Crohns Disease
Keywords: Randomized Controlled Trial; Factorial Design; Fecal Microbial Transplantation; Crohns disease exclusion diet; Crohns disease; Advanced therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fecal microbiota transplantation(FMT) with Crohns disease exclusion diet (CDED) and advanced therapy (Experimental): 1. FMT via colonoscopy at 0, 2 and 6 weeks (preceded by 3 days antibiotics, only before first procedure) followed by (if treatment responder) 8 weekly during maintenance till 42 weeks 2. Crohn disease exclusion diet(CDED) throughout the study 3. Advanced therapy as standard dose and schedule
  Interventions: Other: Fecal Microbial Transplantation; Other: Crohns Disease Exclusion Diet; Other: Advanced therapy
- Fecal microbiota transplantation (FMT) with sham diet and Advanced therapy (Experimental): 1. FMT via colonoscopy at 0, 2 and 6 weeks (preceded by 3 days antibiotics, only before first procedure) followed by (if treatment responder) 8 weekly during maintenance till 42 weeks 2. Dietary counselling throughout the study 3. Advanced therapy as standard dose and schedule
  Interventions: Other: Fecal Microbial Transplantation; Other: Sham Diet; Other: Advanced therapy
- Sham FMT with Crohns disease exclusion diet (CDED) and advanced therapy (Experimental): 1. Sham FMT with instillation of clean water at 0, 2 and 6 weeks (preceded by 3 days antibiotics, only before first procedure) followed by (if treatment responder) - 8- weekly during maintenance till 42 weeks 2. CDED throughout the study 3. Advanced therapy as standard dose and schedule
  Interventions: Other: Crohns Disease Exclusion Diet; Other: Sham transplantation; Other: Advanced therapy
- Sham Diet with Sham FMT with advance therapy (Sham Comparator): 1.Sham FMT with instillation of clean water at 0, 2 and 6 weeks (preceded by 3 days antibiotics, only before first procedure) followed by (if treatment responder) - 8- weekly during maintenance till 42 weeks 2. Dietary counselling throughout the study 3. Advanced therapy as standard dose and schedule.
  Interventions: Other: Sham transplantation; Other: Sham Diet; Other: Advanced therapy

INTERVENTIONS:
Other: Fecal Microbial Transplantation — This will involve colonoscopic instillation of fecal transplant
  Arms: Fecal microbiota transplantation (FMT) with sham diet and Advanced therapy; Fecal microbiota transplantation(FMT) with Crohns disease exclusion diet (CDED) and advanced therapy
Other: Crohns Disease Exclusion Diet — The modified diet plan will be given to each study participant
  Arms: Fecal microbiota transplantation(FMT) with Crohns disease exclusion diet (CDED) and advanced therapy; Sham FMT with Crohns disease exclusion diet (CDED) and advanced therapy
Other: Sham transplantation — Sham transplantation will involve saline infusion via colonoscopy
  Arms: Sham Diet with Sham FMT with advance therapy; Sham FMT with Crohns disease exclusion diet (CDED) and advanced therapy
Other: Sham Diet — Dietary counselling alone
  Arms: Fecal microbiota transplantation (FMT) with sham diet and Advanced therapy; Sham Diet with Sham FMT with advance therapy
Other: Advanced therapy — Advanced therapy as standard dose and schedule

SUMMARY:
Advanced therapies including biologics and small molecules target specific inflammatory pathways. IBD's multifactorial etiology means that blocking a single pathway may not be sufficient for all patients. Even when combination of advanced therapies are used, the incremental benefits often diminish, reflecting the therapeutic ceiling. Furthermore, safety concerns also limit the potential to push beyond this ceiling. Increasing the dose or adding more immunosuppressive agents can lead to a higher risk of infections, malignancies, and other adverse effects, making it impractical to continually intensify treatment. Understanding the therapeutic ceiling in IBD highlights the need for innovative approaches that go beyond current strategies. Given the diverse microbial and immunological landscapes in IBD combining fecal microbiota transplantation (FMT) and Crohn's Disease Exclusion Diet (CDED) with advanced therapies represents a promising approach to break the therapeutic ceiling in CD. This strategy leverages the complementary mechanisms of action of FMT/CDED and advance therapies, potentially offering a more comprehensive treatment modality that addresses the complex and multifactorial nature of IBD. FMT involves the transfer of gut microbiota from a healthy donor to a patient, aiming to restore a balanced microbial community in the intestines. This can help modulate the immune system and reduce inflammation, which are central to Crohn's disease pathology. This study seeks to provide evidence on whether addition of microbiota manipulation by FMT and CDED offers additional benefits when used alongside advance therapies in active CD. The findings from this RCT are expected to significantly enhance treatment strategies, ensuring that patients receive the most effective and appropriate care based on robust scientific evidence. This multi-center double blind placebo-controlled RCT will randomize patients in 1:1:1:1 ratio to FMT, CDED and advance therapy vs sham FMT with advance therapy and CDED vs FMT, Advance therapy and sham diet vs Advance therapy with sham FMT and sham diet for induction and maintenance of remission in patients of active Crohn's disease. Randomization will be held centrally to ensure concealment of allocation. Random numbers will be generated by computerized random number schedule (The RAND), and the randomization list and numbered packing of the intervention will be prepared by a person not involved in the study. Randomization will be performed using permuted blocks of 8. Both the patient and the investigator will be blinded to the intervention

DETAILED DESCRIPTION:
This is a multicenter, double-blind, factorial randomized controlled trial (RCT) evaluating the efficacy of microbiome manipulation strategies in patients with active Crohn's Disease (CD) undergoing advanced therapy (biologics or small molecules). The study will be conducted across six clinical centers in India, with an additional center designated for microbiome analysis.

Randomization and Blinding:

Randomization: Centralized, computer-generated randomization using permuted blocks of 8, 12, and 16 to ensure equal distribution across intervention arms.

Stratification: Not more than 1/3rd patients should be biological therapy exposed

Blinding:

The blinded team includes patients and principal investigators. Endoscopists administering FMT/sham FMT and dietitians providing dietary counseling will be unblinded

Sham-Control Methods:

FMT Sham: Sterile clean water infusions via colonoscopy. Diet Sham: Dietary counseling without any modification

Intervention Arms:

Patients are randomized into one of four treatment groups:

FMT + CDED + Advanced Therapy (Group A) FMT + Sham Diet + Advanced Therapy (Group B) Sham FMT + CDED + Advanced Therapy (Group C) Sham FMT + Sham Diet + Advanced Therapy (Group D)

Fecal Microbiota Transplantation (FMT):

FMT Route: Administered via colonoscopy.

FMT Schedule:

Induction Phase: Weeks 0, 2, and 6. Maintenance Phase: Every 8 weeks (weeks 10, 18, 26, 34, 42) for responders.

Preparation:

Donor Selection: Multi-donor approach with prescreening FMT Processing: 50 g stool freshly prepared and instilled within 4 hours.

Delivery Locations:

Week 0 (Bowel Preparation): Right colon/terminal ileum. Weeks 2 and 6 (No Bowel Preparation): Left colon. Crohn's Disease Exclusion Diet (CDED)

Diet Structure:

Induction Phase (Weeks 0-6): Elimination of specific pro-inflammatory dietary components.

Maintenance Phase (Weeks 6-48): Gradual reintroduction of certain food groups. Monitoring: Adherence tracked using the IBD NutriCare app, diet recall logs, and DietCal software.

Sham Diet: Patients follow a standard healthy diet with general dietary counseling.

Assessments and Data Collection Baseline Assessments (Week 0) Clinical Data: Crohn's Disease Activity Index (CDAI), stool frequency, rectal bleeding, and symptom tracking.

Laboratory Tests:

Hemogram, renal/liver function tests, blood glucose. Inflammatory Markers: C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), fecal calprotectin (FCP).

Microbiome Analysis: Stool samples stored at -80°C for sequencing.

Endoscopic Evaluation:

Scoring: Simple Endoscopic Score for CD (SES-CD). Blinded Central Review: Videos assessed by two independent readers; discrepancies adjudicated by a third reader.

Histology: Biopsies analyzed using DCA score (Distribution Chronicity and Activity).

Follow-up Assessments

Visit Schedule:

Induction Phase: Weeks 2, 4, 6, and 10. Maintenance Phase: Every 8 weeks (weeks 18, 26, 34, 42, and 48). Clinical Assessments: CDAI, PRO2 symptom tracking, medication adherence checks. Endoscopy: Week 10 and Week 48; central scoring of videos. Diet Adherence: Assessed at weeks 2, 4, 6, and 10, then every 8 weeks. Microbiome Sampling: Stool samples collected at weeks 10 and 48. Safety Monitoring and Adverse Events

Adverse Event (AE) Classification:

CTCAE Grading (Grade 1-5) for treatment-related AEs. Serious Adverse Events (SAEs): Hospitalization, life-threatening events, or disability.

Safety Monitoring Plan:

Pre-procedural safety checks for each FMT session. Immediate post-FMT monitoring (48 hours). Late safety assessments (14 days post-FMT, then every visit). Unblinding Procedure: Allowed only for SAE management with DSMB approval. Data Management and Statistical Analysis

Electronic Data Capture (EDC):

Platform: REDCap database with tiered access permissions. Audit Trails: Secure logs of data entry and modification.

Dietary Data Processing:

IBD NutriCare app logs converted into macronutrient composition reports. Adherence scoring based on 80% compliance threshold.

Microbiome Data Processing:

Samples sequenced at IIIT-Delhi, analyzed for diversity indices and metabolic pathways.

Statistical Plan:

Primary Analysis: Intention-to-treat (ITT) and per-protocol (PP) analyses. Longitudinal Modeling: Mixed-effects models for repeated measures.

Effect Size Estimation:

Sample size: 168 patients (42 per arm).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active Crohn disease in whom FMT is feasible
2. Active Crohn's disease who are candidates for advanced therapy (steroid refractory, Immunomodulator intolerant or refractory and moderately severe disease at the time of inclusion) or patients who have an intolerance to or have lost response to advanced therapies must have had their last treatment at least five half-lives prior randomization.
3. Aged between 18-75 years
4. CDAI greater than 150 and/or SES-CD equal or greater than 6 (or equal or greater than 4 if isolated ileal disease)

Exclusion Criteria:

1. Patients in remission (CDAI less than 150)
2. Stricturing disease (non-passable stricture) in whom FMT is not feasible
3. Fistulising phenotype or Perianal fistula or abscess
4. Isolated L4 disease
5. Active TB or Sepsis
6. Pregnant or lactating women
7. Patients with co-morbidities like CAD/CLD/CKD
8. Previous surgery for CD
9. Declining consent or not willing for FMT or diet advice
10. Patients with current or recent history of clinically severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological disease.
11. Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) or positive test for Clostridioides difficile toxin at screening#
12. Patients infected with human immunodeficiency virus (HIV) #The patients with positive assay will be treated appropriately and tests will be repeated.

Those with negative assay and persistent activity will be included in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clinical remission and endoscopic response at week 10 | 10 weeks
  Proportion of patients with clinical remission (defined as CDAI less than 150) and endoscopic response( defined decline in SES-CD by greater than 50%)
Proportion of patients with clinical remission and endoscopic remission at week 10 | 48 weeks
  Proportion of patients with clinical remission (defined as Crohn's disease activity index less than 150) and endoscopic remission (defined as Simple Endoscopic Score for Crohn's disease patients less than 3)

SECONDARY OUTCOMES:
Proportion of patients with clinical response at Week 10 | 10 weeks
  Proportion of patients with clinical response is defined as either CDAI decrease from baseline of at least 70 points or CDAI less than 150
Proportion of patients with PRO2 Remission at Week 10 | 10 weeks
  Proportion of patients with PRO2 Remission which is defined as Abdominal pain subscore of not more than 1 (on a scale of 0-3) and liquid or very soft stool (Bristol stool scale type 6 or 7) frequency subscore of not more than 3 calculated as a mean of 7 day count
Proportion of patients with endoscopic response at Week 10 | 10 weeks
  Proportion of patients with endoscopic response which is defined as 50% reduction from baseline on SES-CD
Fecal microbiome and metabolite signature between responders and non-responders at week 10 | 10 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Proportion of patients with biomarker remission at Week 10 | 10 weeks
  Proportion of patients with biomarker remission which is defined as fecal calprotectin ≤150 mcg/g
Proportion of patients with adverse events at Week 10 | 10 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))
Proportion of patients with clinical response at Week 48 | 48 weeks
  Proportion of patients with clinical response is defined as either CDAI decrease from baseline of at least 70 points or CDAI less than 150
Proportion of patients with PRO2 remission at Week 48 | 48 weeks
  Proportion of patients with PRO2 remission is defined as Abdominal pain subscore of not more than 1 (on a scale of 0-3) and liquid or very soft stool (Bristol stool scale type 6 or 7) frequency subscore of not more than 3 calculated as a mean of 7 day count
Proportion of patients with endoscopic response at Week 48 | 48 weeks
  Proportion of patients with endoscopic response defined as 50% reduction from baseline on SES-CD
Proportion of patients with Endoscopic remission at Week 48 weeks | 48 weeks
  Proportion of patients with Endoscopic remission defined as a SES-CD score of 2 or less
Proportion of patients with corticosteroid-free clinical remission at Week 48 | 48 weeks
  Proportion of patients with corticosteroid-free clinical remission is defined as the CDAI<150 with no exposure to steroids over the previous 8 weeks
Fecal microbiome and metabolite signature between responders and non-responders at Week 48 | 48 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Proportion of patients with biomarker remission at Week 48 | 48 weeks
  Proportion of patients with biomarker remission which is defined as fecal calprotectin ≤150 mcg/g
Proportion of patients with adverse event at Week 48 | 48 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))
Proportion of patients with adverse event at Week 6 | 6 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))
Proportion of Patients Experiencing Adverse Events at Week 26 | 26 weeks
  Proportion of Patients Experiencing Adverse Events (will be assessed according to common criteria for adverse events (CTCEA))

CONTACTS AND LOCATIONS:
Overall Officials: Prof Vineet Ahuja, DM Gastroenterology, Principal Investigator — Department of Gastroenterology, AIIMS, New Delhi
Locations (6):
- India (6):
  - Department of Gastroenterology, Lisie Hospital, Kochi, Kerala
  - Lokmanya Tilak Municipal General Hospital and Lokmanya Tilak Municipal Medical College, Sion, Mumbai, Maharashtra
  - Department of Gastroenterology and Human Nutrition, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Department of Gastroenterology, Dayanand Medical College, Ludhiana, Punjab
  - Department of Gastroenterology, Institute of Medical Sciences, Varanasi, Uttar Pradesh
  - Department of Gastroentrology, Postgraduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No